CLINICAL TRIAL: NCT00081653
Title: Double-blind, Partially Randomized, Parallel Group, Multicenter Study to Assess the Efficacy and Safety of 100 mg and 150 mg Monthly Oral Ibandronate in Women With Postmenopausal Osteoporosis Having Completed the Phase III Oral Ibandronate Trial BM16549
Brief Title: A Study of Bonviva (Ibandronate) in Women With Post-Menopausal Osteoporosis Previously Treated With Bonviva
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA17903
Record Dates: First submitted 2004-04-19; First posted 2004-04-21 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Post-Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Active Comparator)
  Interventions: Drug: ibandronate [Bonviva/Boniva]

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 3 years
  Arms: 1
Drug: ibandronate [Bonviva/Boniva] — 100mg po monthly for 3 years
  Arms: 2

SUMMARY:
This 2 arm study will assess the long-term efficacy and safety of oral treatment with 100mg or 150mg Bonviva in women with post-menopausal osteoporosis who have previously completed Bonviva study BM16549 (MOBILE study). Patients will receive Bonviva either 100mg po monthly, or 150mg po monthly. Patients will also receive daily supplementation with vitamin D and calcium. The anticipated time of study treatment is 2+ years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* successful completion of Bonviva study BM16549, with at least 75% compliance;
* ambulatory.

Exclusion Criteria:

* malignant disease diagnosed within the previous 12 years (except basal cell cancer that has been successfully removed);
* breast cancer diagnosed within the previous 22 years.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2004-05; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (5):
  - Loma Linda, California
  - Lakewood, Colorado
  - Omaha, Nebraska
  - Livingston, New Jersey
  - Portland, Oregon
- Belgium (2):
  - Liège
  - Merksem
- São Paulo, Brazil
- Czechia (2):
  - Pilsen
  - Prague
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Lyon, France
- Germany (2):
  - Berlin
  - Hanover
- Hungary (4):
  - Balatonfüred
  - Budapest
  - Kiskunhalas
  - Zalaegerszeg
- Siena, Italy
- Mexico (2):
  - León
  - Obregón
- Norway (2):
  - Haugesund
  - Stavanger
- Poland (2):
  - Krakow
  - Warsaw
- Spain (2):
  - Barcelona
  - Madrid
- Southampton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 31 centers over the period of 18 May 2004 to 28 November 2007.
Pre-assignment Details: Eligible for the study were patients having completed Study BM16549 (NCT00081653) and who had complied with the monthly regimen for 75 percent (%) or more.
Groups:
- Ibandronate 100 Milligrams (mg): 100 mg ibandronate oral (PO) monthly and monthly oral placebo (corresponding to the 150 mg tablet)
- Ibandronate 150 mg: 150 mg ibandronate PO monthly and monthly oral placebo (corresponding to the 100 mg tablet)
Period: Overall Study
Arm/Group | Ibandronate 100 Milligrams (mg) | Ibandronate 150 mg
Started | 358 (Patients entering Study MA17903 from Study BM16549) | 361 (Patients entering Study MA17903 from Study BM16549)
Completed | 311 (Completed 3 years of treatment) | 324 (Completed 3 years of treatment)
Not Completed | 47 | 37
Not completed — Adverse Event | 23 | 17
Not completed — Lost to Follow-up | 2 | 4
Not completed — Refused Treatment | 18 | 14
Not completed — Low bone mineral density | 1 | 0
Not completed — Bone loss | 2 | 0
Not completed — Participant leaving country | 1 | 0
Not completed — Loss of bone mass | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent -To - Treat (ITT) population: All participants who were randomized into this study, received at least one dose of the trial medication, and had at least one follow-up efficacy data point (BMD or serum C-terminal peptide cross-links of Collagen Type I [CTX]).
Groups:
- Ibandronate 100 mg: 100 mg ibandronate PO monthly and monthly oral placebo (corresponding to the 150 mg tablet)
- Total: Total of all reporting groups
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg | Total
Number analyzed (Participants) | 358 | 361 | 719
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (6.55) | 67.7 (6.8) | 67.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 358 | 361 | 719
  Male | 0 | 0 | 0
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.87 (4.957) | 26.04 (3.976) | 25.96 (4.489)
Race, Customized [Number; unit: participants]
  Caucasian/White | 341 | 338 | 679
  Black | 0 | 1 | 1
  Oriental | 0 | 1 | 1
  Hispanic | 17 | 20 | 37
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Absolute Change From Baseline in Mean Total Hip BMD
Description: BMD was measured by a single DXA scan of the hip. Scores between -1 and -2.5 indicate Osteopenia (thin bones). Less than -2.5 indicate Osteoporosis (porous bones).
Time Frame: Baseline and 12, 24 and 36 months
Population: ITT Population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 347 | 348
g/cm^2
  Baseline (n=345,348) | 0.7680 (0.1093) | 0.7862 (0.1112)
  Month 12 (n=347,346) | 0.7669 (0.1097) | 0.7888 (0.1116)
  Change from Baseline at Month 12 (n=344,345) | -0.0004 (0.0204) | 0.0025 (0.0200)
  Month 24 (n=322,336) | 0.7686 (0.1104) | 0.7882 (0.1124)
  Change from Baseline at Month 24 (n=319,335) | -0.0010 (0.0227) | 0.0031 (0.0214)
  Month 36 (n=301,321) | 0.7663 (0.1133) | 0.7834 (0.1128)
  Change from Baseline at Month 36 (n=298,320) | -0.0061 (0.0254) | -0.0030 (0.0252)

2. Secondary Outcome: Relative Percent Change From Baseline in Mean Total Hip BMD
Description: as for outcome 1
Time Frame: Baseline, 12, 24 and 36 months
Population: ITT Population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 344 | 345
percent change in BMD
  Change from Baseline at Month 12 (n=344,345) | -0.0169 (2.8582) | 0.3459 (2.5849)
  Change from Baseline at Month 24 (n=319,335) | -0.1092 (3.1040) | 0.4378 (2.8062)
  Change from Baseline at Month 36 (n=298,320) | -0.8045 (3.3448) | -0.3496 (3.3254)

3. Secondary Outcome: Absolute Change From Baseline of Trough Serum CTX
Description: CTX is a measure of bone resorption and is measured as ng/mL. Blood samples for the Month 6 values were collected 6 days after the 6-month dose; therefore, the Month 6 values are not true 'trough' values.
Time Frame: Baseline, 6, 12, 24 and 36 months
Population: ITT population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 57 | 68
ng/mL
  Baseline (n= 56,68) | 0.232 (0.1520) | 0.219 (0.1799)
  Month 6 Postdose (n=56,68) | 0.176 (0.1826) | 0.126 (0.1222)
  Change from Baseline at Month 6 Postdose (n=55,67) | -0.055 (0.1307) | -0.093 (0.1510)
  Month 12 (n=57,67) | 0.279 (0.1617) | 0.208 (0.1073)
  Change from Baseline at Month 12 (n=56,67) | 0.048 (0.1303) | -0.011 (0.1406)
  Month 24 (n=54,65) | 0.309 (0.1406) | 0.266 (0.1548)
  Change from Baseline at Month 24 (n=53,65) | 0.088 (0.1203) | 0.048 (0.1607)
  Month 36 (n=51,60) | 0.410 (0.1805) | 0.380 (0.2036)
  Change from Baseline at Month 12 (n=50,60) | 0.205 (0.1396) | 0.174 (0.1549)

4. Primary Outcome: Absolute Change From Baseline in Mean Lumbar Spine (L2 - L4) BMD
Description: Absolute change from Baseline in mean BMD of the lumbar spine (L2 - L4) measured as grams per square centimeter (g/cm^2). This was baseline of Study MA17903 after two years of treatment in the core study (BM16549 [NCT00081653]).
Time Frame: Baseline and Months 12, 24 and 36
Population: ITT population; number (n) equals (=) number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 347 | 346
g/cm^2
  Baseline (n=347,346) | 0.7916 (0.0814) | 0.7977 (0.0791)
  Month 12 (n=347,346) | 0.7977 (0.0831) | 0.8069 (0.0819)
  Change from Baseline at Month 12 (n=346,343) | 0.0061 (0.0293) | 0.0097 (0.0289)
  Month 24 (n=323,336) | 0.8048 (0.0861) | 0.8111 (0.0852)
  Change from Baseline at Month 24 (n=322,333) | 0.0131 (0.0332) | 0.0140 (0.0356)
  Month 36 (n=308,320) | 0.8090 (0.0916) | 0.8155 (0.0892)
  Change from Baseline at Month 36 (n=307, 318) | 0.0172 (0.0382) | 0.0194 (0.0383)

5. Primary Outcome: Relative Percent (%) Change From Baseline in Mean Lumbar Spine (L2 - L4) Bone Mineral Density (BMD)
Description: BMD was measured by a single dual-energy X-ray absorptiometry (DXA) scan of the lumbar spine (BMD of at least 2 vertebrae [L2-L4] that were not fractured and not affected by osteoarthritis to such a degree that BMD measurement would be compromised) at the time of enrollment and at Months 12, 24 and 36. This was baseline of Study MA17903 after two years of treatment in the core study (BM16549 [NCT00081653]).
Time Frame: Baseline and Months 12, 24 and 36
Population: ITT population: n = number of participants analyzed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 346 | 343
percent change
  Change from Baseline at Month 12 (n=346,343) | 0.8348 (3.8118) | 1.2550 (3.6402)
  Change from Baseline at Month 24 (n=322,333) | 1.6921 (4.2385) | 1.7865 (4.5058)
  Change from Baseline at Month 36 (n=307,318) | 2.1794 (4.9176) | 2.4322 (4.8146)

6. Secondary Outcome: Relative Percent Change From Baseline of Trough Serum CTX
Description: CTX is a measure of bone resorption and is measured as nanograms per milliliter (ng/mL). Blood samples for the Month 6 values were collected 6 days after the 6-month dose; therefore, the Month 6 values are not true 'trough' values.
Time Frame: Baseline, 6,12, 24 and 36 months
Population: ITT population; n = number of participants analyzed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Ibandronate 100 mg: 100 mg ibandgronate PO monthly and monthly oral placebo (corresponding to the 150 mg tablet)
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg
Number analyzed (Participants) | 56 | 68
percent change
  Baseline (n=56,68) | 0.232 (0.1520) | 0.219 (0.1799)
  Month 6 Postdose (n=56, 67) | 0.176 (0.1826) | 33.109 (40.3544)
  Change from Baseline at Month 6 Postdose (n=55,67) | -24.622 (43.4212) | -33.109 (40.3544)
  Month 12 (n=57,67) | 0.279 (0.1617) | 0.208 (0.1073)
  Change from Baseline at Month 12 (n=56,67) | 31.121 (58.9832) | 25.125 (86.5607)
  Month 24 (n=54,65) | 0.309 (0.1406) | 0.266 (0.1548)
  Change from Baseline at Month 24 (n=53,65) | 58.657 (65.3128) | 53.704 (74.9810)
  Month 36 (51,60) | 0.410 (0.1805) | 0.380 (0.2036)
  Change from Baseline at Month 36 (n=50,60) | 121.106 (97.9878) | 138.502 (125.7590)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of informed consent until 15 days after the final visit at 36 months.
Arm/Group | Ibandronate 100 mg | Ibandronate 150 mg
Serious Adverse Events (participants affected / at risk) | 68/358 | 70/361
Other Adverse Events (participants affected / at risk) | 187/358 | 185/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 100 mg (N=358) | Ibandronate 150 mg (N=361)
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 4
Wrist fracture (Injury, poisoning and procedural complications) | 3 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 3
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 1
Angina pectoris (Cardiac disorders) | 0 | 5
Myocardial Ischaemia (Cardiac disorders) | 2 | 1
Aortic valve stenosis (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac fibrillation (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritoneal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tetanus (Infections and infestations) | 0 | 1
Ureteritis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 0 | 2
Intermittent claudication (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Cataract (Eye disorders) | 3 | 2
Keratoconus (Eye disorders) | 0 | 1
Entropion (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 3
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Cervix disorder (Reproductive system and breast disorders) | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Vaginal disorder (Reproductive system and breast disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Central obesity (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Diabetes mellitus management (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 100 mg (N=358) | Ibandronate 150 mg (N=361)
Nasopharyngitis (Infections and infestations) | 46 | 40
Urinary tract infection (Infections and infestations) | 22 | 27
Bronchitis (Infections and infestations) | 24 | 21
Influenza (Infections and infestations) | 22 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 36
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 15
Hypertension (Vascular disorders) | 42 | 49
Hypercholesterolaemia (Metabolism and nutrition disorders) | 30 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No